CLINICAL TRIAL: NCT05653700
Title: Atrium Health - Arena Labs Research Protocol
Brief Title: Arena Labs - Improving Clinician Well Being
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00090882
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Results first posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2023-08

CONDITIONS: Mental Health Disorder
Keywords: professional fulfillment; physiological resilience; high-stress environment
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study is a prospective randomized controlled longitudinal crossover design with a per protocol analysis integrating one sensor (WHOOP, inc Platform) and one educational intervention (Arena Strive Platform).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arena Strive (Experimental): The experimental intervention employed in this study will be a 12-week, multi-phased approach involving an asynchronous learning and coaching experience (6 weeks), and exploration phase (6 weeks).
  Interventions: Device: Arena Strive
- Control Cohort (Other): Participants randomized into the control cohort - survey at baseline and end of the study
  Interventions: Other: Control Cohort

INTERVENTIONS:
Device: Arena Strive — This second-generation platform provides frontline clinicians with a comprehensive journey to access the tools, training, and technology used by other high-pressure fields to increase performance and enhance resilience. The experimental intervention employed in this study will be a 12-week, multi-phased approach involving an asynchronous learning and coaching experience (6 weeks), and exploration phase (6 weeks).
  Arms: Arena Strive
Other: Control Cohort — Participants randomized into the control cohort - survey at baseline and end of the study
  Arms: Control Cohort

SUMMARY:
To determine the efficacy of the asynchronous performance coaching platform, Arena Strive at changing measures of physiological resilience, professional fulfillment, burnout, and self-valuation in full time clinicians.

DETAILED DESCRIPTION:
This study is a prospective randomized controlled longitudinal crossover design with a per protocol analysis integrating one sensor (WHOOP, inc Platform) and one educational intervention (Arena Strive Platform). The WHOOP sensor collects data on heart rate (HR), heart rate variability (HRV), and sleep data, and will be worn by all participants in the experimental intervention. Participants will be asked to wear the biometric sensor for 12 weeks but will have optional access to the device for a total of 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Employed full time by an Atrium Health affiliated entity
* Age 18+
* Willing and able to give written informed consent for study participation
* Healthcare workers working ≥ 36 hours of clinical duties/week
* Willingness to wear WHOOP and keep it charged for the entire duration of study
* Have a smart phone for pairing with WHOOP and the Arena Strive platform

Exclusion Criteria:

* Current diagnosis of a sleep-related breathing disorder including obstructive sleep apnea not being treated (with or without continuous positive airway pressure (CPAP) treatment)
* Circadian rhythm sleep-wake disorders
* Narcolepsy
* Recurrent isolated sleep paralysis
* Restless legs syndrome
* Periodic Leg Movement Disorder
* Comorbid nocturia or other conditions (benign prostatic hyperplasia) resulting in frequent need to get out of bed to use the bathroom during the night (≥3 times per night average)
* Atrial Fibrillation
* Chronic obstructive pulmonary disease (COPD) other than mild, pulmonary fibrosis or severe chronic lung disease
* Sleep apnea or undergoing treatment for a sleep related illness
* Lack of availability of iPhone or Android device

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-03-16 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Lobdell, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Sanger Heart and Vascular Institute, Charlotte, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (test, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified or this purpose

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Non Response is difference in Subject numbers
Groups:
- Arena Strive: The experimental intervention employed in this study will be a 12-week, multi-phased approach involving an asynchronous learning and coaching experience (6 weeks), and exploration phase (6 weeks). All participants will receive a Whoop device to capture biometric data.
  WHOOP Sensor: The WHOOP sensor collects data on heart rate (HR), heart rate variability (HRV), and sleep data
  Arena Strive: This second-generation platform provides frontline clinicians with a comprehensive journey to access the tools, training, and technology used by other high-pressure fields to increase performance and enhance resilience.
- Control Cohort: Participants randomized into the control cohort - the intervention is the survey at baseline, mid-point, and end of the study
Period: Overall Study
Arm/Group | Arena Strive | Control Cohort
Started | 29 | 14
Completed | 20 | 14
Not Completed | 9 | 0
Not completed — Non Responders | 9 | 0

BASELINE CHARACTERISTICS:
Population: Patients were randomized into either control or intervention group (Arena Strive)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arena Strive | Control Cohort | Total
Number analyzed (Participants) | 29 | 14 | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 14 | 43
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Measurement was not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Change in Heart Rate Variability
Description: measured by the WHOOP biometric device - The WHOOP wearable brings hi-tech features including sleep, workout, heart rate feedback and more advanced biometrics in a simple package - the latest, most advanced fitness and health wearable available. Monitor your recovery, sleep, training, and health, with personalized recommendations and coaching feedback. Values represent heart rate at specific intervals. The higher the HRV generally the better
Time Frame: Week 16
Population: non response
Measure: Mean (95% Confidence Interval); unit: Milliseconds
Groups:
- Arena Strive: The experimental intervention employed in this study will be a 12-week, multi-phased approach involving an asynchronous learning and coaching experience (6 weeks), and exploration phase (6 weeks).
  Arena Strive: This second-generation platform provides frontline clinicians with a comprehensive journey to access the tools, training, and technology used by other high-pressure fields to increase performance and enhance resilience.
Arm/Group | Arena Strive
Number analyzed (Participants) | 29
Milliseconds
  Beginning (Week 6) | 39 [27 to 56]
  Mid (Week 12) | 47 [32 to 65]
  End (Week 16) | 54 [35 to 82]

2. Primary Outcome: Change in Resting Heart Rate
Description: measured by the WHOOP biometric device - The WHOOP wearable brings hi-tech features including sleep, workout, heart rate feedback and more advanced biometrics in a simple package - the latest, most advanced fitness and health wearable available. Monitor your recovery, sleep, training, and health, with personalized recommendations and coaching feedback. The lower heart rate at rest implies more efficient heart function and better cardiovascular fitness.
Time Frame: Week 16
Population: non response
Measure: Mean (95% Confidence Interval); unit: Beats per Minute
Arm/Group | Arena Strive
Number analyzed (Participants) | 29
Beats per Minute
  Beginning (Week 6) | 63 [57 to 68]
  Mid (Week 12) | 60 [55 to 65]
  End (Week 16) | 57 [51 to 61]

3. Primary Outcome: Change in Time Spent in Bed
Description: measured by the WHOOP biometric device - The WHOOP wearable brings hi-tech features including sleep, workout, heart rate feedback and more advanced biometrics in a simple package - the latest, most advanced fitness and health wearable available. Monitor your recovery, sleep, training, and health, with personalized recommendations and coaching feedback.
Time Frame: Week 16
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Arena Strive
Number analyzed (Participants) | 29
hours
  Beginning (Week 6) | 7.69 [6.83 to 8.67]
  Mid (Week 12) | 7.60 [6.60 to 8.55]
  End (Week 16) | 7.59 [6.56 to 9.05]

4. Primary Outcome: Change in Sleep Quality
Description: as for outcome 3
Time Frame: Week 16
Population: Data not collected
Arm/Group | Arena Strive
Number analyzed (Participants) | 0

5. Primary Outcome: Change in Sleep Consistency
Description: as for outcome 3
Time Frame: Week 16
Population: Data not collected
Arm/Group | Arena Strive
Number analyzed (Participants) | 0

6. Primary Outcome: Change in Sleep Debt
Description: as for outcome 3
Time Frame: Week 16
Population: Data not collected
Arm/Group | Arena Strive
Number analyzed (Participants) | 0

7. Primary Outcome: Change in Amount of Burn Out (MBI) Malasch Burnout Inventory
Description: Each item is measured on a scale of 0 to 6 and Total scores range from 0 (less/better burnout) - to 42 (more/worse burnout) - Total score of 17 or less: low level burnout total between 18 and 29 inclusive: moderate burnout total over 30: high-level of burnout
Time Frame: Week 16
Population: difference in Subject number due to Non-Responders
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control Cohort: Participants randomized into the control cohort - the intervention is the survey at baseline and end of the study
Arm/Group | Arena Strive | Control Cohort
Number analyzed (Participants) | 29 | 14
score on a scale
  Week 6: number analyzed (Participants) | 28 | 14
  Week 6 | 20 (9) | 22 (9)
  Week 12: number analyzed (Participants) | 26 | 13
  Week 12 | 17 (8) | 15 (10)
  Week 16: number analyzed (Participants) | 20 | 14
  Week 16 | 16 (10) | 32 (6)

8. Primary Outcome: Change in Self-reported Professional Fulfillment (PFI)
Description: collected by means of a survey link at key benchmark moments throughout the intervention period - Each item within PFI scored from 0 to 4 with higher scores being more favorable - scores range from 0 - 24 with higher scores denoting higher fulfillment
Time Frame: Week 16
Population: Survey non response accounts for difference in number of Subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arena Strive | Control Cohort
Number analyzed (Participants) | 29 | 14
score on a scale
  Week 6 | 2.30 (0.75) | 2.50 (0.73)
  Week 12: number analyzed (Participants) | 26 | 13
  Week 12 | 2.58 (0.67) | 2.14 (0.73)
  Week 16: number analyzed (Participants) | 20 | 14
  Week 16 | 2.69 (0.99) | 2.07 (0.74)

9. Primary Outcome: Change in Self-valuation Scores (Stanford Self-Vaulation)
Description: collected by means of an in-app survey at key benchmark moments throughout the intervention period - Each item in the self-valuation scale included 4 items measured on a 5-point (0-4) Likert scale lower scores meaning more positivity -scores range from 0 - 16 with lower score denoting more positivity
Time Frame: Week 16
Population: Survey non response accounts for difference in Subject number
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arena Strive | Control Cohort
Number analyzed (Participants) | 29 | 14
score on a scale
  Week 6 | 5.93 (2.42) | 6.57 (2.59)
  Week 12: number analyzed (Participants) | 26 | 13
  Week 12 | 7.19 (2.84) | 6.85 (2.70)
  Week 16: number analyzed (Participants) | 20 | 14
  Week 16 | 7.60 (2.68) | 7.64 (2.87)

10. Primary Outcome: Change in Personal Achievement (MBI)
Description: "Each Item Measured on a scale of 0 to 6; Total 33 or less: high-level burnout - Total between 34 and 39 inclusive: moderate burnout - Total greater than 40: low-level burnout" Scores range from 0 - 48 with higher scores denoting less burnout
Time Frame: week 16
Population: difference in Subject number due to non responders
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arena Strive | Control Cohort
Number analyzed (Participants) | 28 | 14
score on a scale
  Week 6 | 38 (8) | 35 (7)
  Week 12: number analyzed (Participants) | 26 | 13
  Week 12 | 37 (9) | 34 (7)
  Week 16: number analyzed (Participants) | 20 | 14
  Week 16 | 37 (9) | 32 (6)

11. Primary Outcome: Change in Depersonalization (MBI)
Description: "Each item measured on a scale of 0 to 6; total score of 5 or less: low level burnout - total between 6 and 11 inclusive: moderate burnout - total over 12 and greater: high-level of burnout" - scores ranging from 0 - 42 with higher scores denoting more burnout
Time Frame: week 16
Population: change in Subject number due to non responders
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arena Strive | Control Cohort
Number analyzed (Participants) | 28 | 14
score on a scale
  Week 6 | 15 (8) | 12 (8)
  week 12: number analyzed (Participants) | 26 | 13
  week 12 | 11 (7) | 14 (9)
  Week 16: number analyzed (Participants) | 20 | 14
  Week 16 | 11 (8) | 15 (10)

12. Primary Outcome: Change in Burnout Scores (PFI) - Professional Fulfillment Index
Description: Scores ranging 0 - 40 with higher scores denoting more exhaustion Likert scale ranging from "not at all" to "extremely" for work exhaustion and interpersonal disengagement item" - lower scores meaning less exhaustion
Time Frame: week 16
Population: change in Subject number due to non responders
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Arena Strive | Control Cohort
Number analyzed (Participants) | 29 | 14
score on a scale
  Week 6 | 1.54 (0.67) | 1.56 (0.55)
  Week 12: number analyzed (Participants) | 26 | 13
  Week 12 | 1.23 (0.63) | 1.76 (0.63)
  Week 16: number analyzed (Participants) | 20 | 14
  Week 16 | 1.20 (0.84) | 1.76 (0.70)

13. Secondary Outcome: Change in Self-reported Satisfaction of the Arena Strive Platform
Description: collected by means of an in-app survey at key benchmark moments throughout the intervention period - client satisfaction questionnaire 8 (CSQ-8) - Scores therefore range from 8 to 32, with higher values indicating higher satisfaction.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Arena Strive: The experimental intervention employed in this study will be a 12-week, multi-phased approach involving an asynchronous learning and coaching experience (6 weeks), and exploration phase (6 weeks).
  Arena Strive: This second-generation platform provides frontline clinicians with a comprehensive journey to access the tools, training, and technology used by other high-pressure fields to increase performance and enhance resilience. WHOOP Sensor: The WHOOP sensor collects data on heart rate (HR), heart rate variability (HRV), and sleep data
Arm/Group | Arena Strive
Number analyzed (Participants) | 22
score on a scale | 25.77 (5.45)

14. Secondary Outcome: Recommendation Score of the Arena Strive Platform
Description: Net Promoter Score with the question of likelihood to recommend - Net Promoter Score (NPS) is calculated by (promoters-detractors)/total respondents. The range is -100 to 100. The closer you are to 100 the more likely recommend.
Time Frame: Week 12
Population: change is Subject number due to non-responses
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arena Strive
Number analyzed (Participants) | 22
score on a scale | 7.45 (2.61)

ADVERSE EVENTS:
Time Frame: through study completion, an average of 16 weeks
Arm/Group | Arena Strive | Control Cohort
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/14
Other Adverse Events (participants affected / at risk) | 0/29 | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05653700/Prot_SAP_001.pdf
  • Informed Consent Form (2023-03-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT05653700/ICF_000.pdf